CLINICAL TRIAL: NCT00592475
Title: A Phase 2, Randomized, Double Blind, Placebo Controlled, Dose Escalation Study to Assess the Safety and Effects of Intravenous Conivaptan on the Hepatic Hemodynamic Response in Stable Euvolemic or Hypervolemic Cirrhotic Patients
Brief Title: A Study to Assess the Safety and Effects of Intravenous (IV) Conivaptan on the Hepatic Hemodynamic Response in Cirrhotic Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cumberland Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 087-CL-089; 2007-001661-15 (EudraCT Number)
Record Dates: First submitted 2008-01-02; First posted 2008-01-14 (Estimated); Results first posted 2010-09-28 (Estimated); Last update posted 2014-05-15 (Estimated); Status verified 2014-04

CONDITIONS: Liver Cirrhosis
Keywords: conivaptan; Liver Cirrhosis; Hypertension, Portal
MeSH Terms: conditions — Liver Cirrhosis; Hypertension, Portal | interventions — conivaptan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Regimen 1 Conivaptan 12.5 mg (Experimental): Conivaptan intravenous loading dose (10 mg) + 2.5 mg continuous infusion over 6.5 hours
  Interventions: Drug: conivaptan
- Regimen 2 Conivaptan 25 mg (Experimental): Conivaptan intravenous loading dose (20 mg) + 5 mg continuous infusion over 6.5 hours
  Interventions: Drug: conivaptan
- Regimen 3 Placebo (Placebo Comparator): Placebo continuous intravenous infusion over 6.5 hours
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: conivaptan — IV
  Arms: Regimen 1 Conivaptan 12.5 mg; Regimen 2 Conivaptan 25 mg
Drug: Placebo — IV
  Arms: Regimen 3 Placebo

SUMMARY:
To evaluate the safety of IV conivaptan in stable euvolemic or hypervolemic cirrhotic patients, and to characterize the effects of IV conivaptan on the hepatic hemodynamic response in patients with cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Institutional Review Board (IRB)/Independent Ethics Committee (IEC)-approved written Informed Consent and appropriate privacy language as per national regulations must be obtained from the subject or legally authorized representative prior to any study-related procedures (including withdrawal of prohibited medication, if applicable)
* Subject is euvolemic or hypervolemic (edematous) secondary to cirrhosis
* Subject has clinical evidence of portal hypertension by the presence of esophageal varices, ascites or both

Exclusion Criteria:

* Clinical evidence of volume depletion or dehydration
* Subject has a history of bleeding from esophageal varices within three months before the start of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-12; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Art Wheeler, MD, Study Director — Cumberland Pharmaceuticals, Inc.
Locations (1):
- Barcelona, Spain

REFERENCES:
- See also: (Link to Prescribing Information) — http://www.astellas.us/docs/vaprisol.pdf

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Regimen 1 Conivaptan 12.5 mg | Regimen 2 Conivaptan 25 mg | Regimen 3 Placebo
Started | 6 | 9 | 5
Completed | 6 | 9 | 5
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Regimen 1 Conivaptan 12.5 mg | Regimen 2 Conivaptan 25 mg | Regimen 3 Placebo | Total
Number analyzed (Participants) | 6 | 9 | 5 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.7 (8.52) | 60.0 (9.72) | 55.2 (7.19) | 59.9 (8.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 0 | 5
  Male | 3 | 7 | 5 | 15
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 6 | 9 | 5 | 20
Underlying Cause of Hyponatremia [Number; unit: Participants] — Patients in the "Not hyponatremia" categories had serum sodium levels of 135-140mEq/L.
  Patients in the "Other" categories had Diuretic treatment.
  Participants
    Euvolemic - Cirrhosis | 1 | 1 | 1 | 3
    Euvolemic - Not Hyponatremia | 2 | 1 | 1 | 4
    Euvolemic - Other | 1 | 0 | 0 | 1
    Hypervolemic - Cirrhosis | 2 | 3 | 3 | 8
    Hypervolemic - Not Hyponatremia | 0 | 3 | 0 | 3
    Hypervolemic - Other | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hepatic Venous Pressure Gradient (HVPG) at 0.5, 1, and 1.5 Hours Post Dose
Description: Change from baseline is calculated as time point minus baseline.
  Baseline procedures were performed prior to study drug administration.
Time Frame: Baseline and 0.5, 1, and 1.5 hours post dose
Population: Participants Analyzed represents Full Analysis Set (FAS): All randomized patients who had at least 1 dose of study drug & who had hepatic venous pressure gradient data at baseline.
  The number of participants per arm is consistent for all categories of the data table.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Regimen 1 Conivaptan 12.5 mg | Regimen 2 Conivaptan 25 mg | Regimen 3 Placebo
Number analyzed (Participants) | 6 | 9 | 5
mmHg
  Baseline | 16.58 (4.375) | 18.33 (4.750) | 15.80 (6.601)
  Change at 0.5 Hours | 0.33 (1.080) | 0.11 (1.318) | -0.10 (0.224)
  Change at 1 Hour | 0.50 (1.844) | 0.56 (1.357) | -0.60 (0.418)
  Change at 1.5 Hours | 0.83 (2.113) | 0.83 (1.732) | -0.10 (1.294)

2. Primary Outcome: Change From Baseline in Hepatic Blood Flow (HBF) at 0.5, 1, and 1.5 Hours Post Dose
Description: as for outcome 1
Time Frame: Baseline and 0.5, 1, and 1.5 hours post dose
Population: Participants Analyzed represents FAS: All randomized patients who had at least 1 dose of study drug & who had hepatic venous pressure gradient data at baseline. (Note: 2 patients were not included in the analysis due to protocol deviations.) The number of participants included in the calculation for each timepoint is noted in the category title.
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Regimen 1 Conivaptan 12.5 mg | Regimen 2 Conivaptan 25 mg | Regimen 3 Placebo
Number analyzed (Participants) | 6 | 9 | 5
mL/min
  Baseline (N= 4; 9; 5) | 581.0 (77.49) | 1182.2 (530.56) | 649.6 (300.44)
  Change at 0.5 Hours (N= 4; 9; 5) | 53.5 (161.30) | -74.1 (558.58) | 73.8 (196.75)
  Change at 1 Hour (N= 4; 9; 4) | 1.3 (160.23) | -70.0 (318.35) | -67.5 (270.27)
  Change at 1.5 Hours (N= 4; 9; 5) | 15.8 (60.26) | -96.0 (390.96) | 40.8 (154.33)

3. Primary Outcome: Change From Baseline in Hepatic Mean Arterial Pressure (MAP) at 0.5, 1, and 1.5 Hours Post Dose
Description: as for outcome 1
Time Frame: Baseline and 0.5, 1, and 1.5 hours post dose
Population: Participants Analyzed represents FAS: All randomized patients who had at least 1 dose of study drug & who had hepatic venous pressure gradient data at baseline.
  The number of participants included in the calculation for each timepoint is noted in the category title.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Regimen 1 Conivaptan 12.5 mg | Regimen 2 Conivaptan 25 mg | Regimen 3 Placebo
Number analyzed (Participants) | 6 | 9 | 5
mmHg
  Baseline (N= 6; 9; 5) | 88.3 (11.89) | 90.3 (7.79) | 84.6 (13.63)
  Change at 0.5 Hours (N= 6; 8; 5) | -6.2 (9.66) | 3.6 (9.97) | 2.6 (4.72)
  Change at 1.0 Hour (N= 6; 9; 5) | -4.2 (9.28) | 5.7 (13.18) | 7.8 (10.92)
  Change at 1.5 Hours (N= 6; 9; 5) | 0 (7.77) | 8.8 (11.39) | 3.4 (6.31)

4. Primary Outcome: Change From Baseline in Blood Pressure at 0.5, 1, 1.5, 2.5, 3.5, 4.5, 5.5, 6.5, 9, 12, and 24 Hours, and Day 8 Post Dose
Description: as for outcome 1
Time Frame: Baseline and 0.5, 1, 1.5, 2.5, 3.5, 4.5, 5.5, 6.5, 9, 12, and 24 hours, and Day 8 post dose
Population: Population is Safety Analysis Set (SAF): All randomized patients who received at least one dose of study medication.
  The number of participants per arm is consistent for all categories of the data table.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Regimen 1 Conivaptan 12.5 mg | Regimen 2 Conivaptan 25 mg | Regimen 3 Placebo
Number analyzed (Participants) | 6 | 9 | 5
mmHg
  Systolic Blood Pressure- Baseline | 112.2 (13.73) | 115.0 (14.42) | 112.8 (12.03)
  Systolic Blood Pressure- Change at 0.5 Hours | 5.3 (13.29) | 5.2 (9.86) | 12.8 (17.54)
  Systolic Blood Pressure- Change at 1 Hour | 5.5 (17.62) | 13.9 (14.12) | 6.8 (21.39)
  Systolic Blood Pressure- Change at 1.5 Hours | 7.8 (20.90) | 7.2 (12.59) | 1.2 (16.27)
  Systolic Blood Pressure- Change at 2.5 Hours | -2.5 (9.65) | -3.8 (8.15) | -2.6 (18.69)
  Systolic Blood Pressure- Change at 3.5 Hours | -6.0 (8.94) | -6.3 (14.83) | -11.4 (10.36)
  Systolic Blood Pressure- Change at 4.5 Hours | -6.2 (12.91) | -17.1 (11.54) | -8.2 (2.95)
  Systolic Blood Pressure- Change at 5.5 Hours | -6.3 (7.20) | -8.7 (14.94) | -7.6 (2.30)
  Systolic Blood Pressure- Change at 6.5 Hours | -8.8 (10.65) | -9.7 (7.73) | -9.4 (15.47)
  Systolic Blood Pressure- Change at 9 Hours | -5.5 (15.35) | 1.9 (11.46) | -7.2 (12.38)
  Systolic Blood Pressure- Change at 12 Hours | -14.0 (21.48) | -7.8 (15.97) | -5.8 (19.41)
  Systolic Blood Pressure- Change at 24 Hours | -10.8 (15.21) | -7.8 (12.53) | -11.0 (5.00)
  Systolic Blood Pressure- Change at 8 Days | -11.5 (7.87) | -7.8 (10.87) | -5.4 (8.41)
  Diastolic Blood Pressure- Baseline | 60.3 (10.65) | 66.3 (9.10) | 71.6 (8.11)
  Diastolic Blood Pressure- Change at 0.5 Hours | 4.5 (3.27) | 4.9 (6.83) | 1.8 (6.10)
  Diastolic Blood Pressure- Change at 1 Hour | 7.3 (5.57) | 5.1 (6.45) | 3.6 (9.84)
  Diastolic Blood Pressure- Change at 1.5 Hours | 9.2 (5.04) | 5.7 (7.04) | 4.0 (11.98)
  Diastolic Blood Pressure- Change at 2.5 Hours | 2.2 (4.83) | -2.1 (6.21) | -3.2 (12.26)
  Diastolic Blood Pressure- Change at 3.5 Hours | 1.0 (2.28) | -0.9 (12.00) | -6.8 (5.54)
  Diastolic Blood Pressure- Change at 4.5 Hours | -2.5 (3.27) | -6.3 (7.45) | -6.4 (7.54)
  Diastolic Blood Pressure- Change at 5.5 Hours | 2.7 (3.93) | -4.2 (7.79) | -9.8 (10.03)
  Diastolic Blood Pressure- Change at 6.5 Hours | -1.0 (7.13) | -4.7 (6.20) | -7.6 (11.01)
  Diastolic Blood Pressure- Change at 9 Hours | 5.0 (5.62) | 0.3 (4.82) | -4.4 (10.01)
  Diastolic Blood Pressure- Change at 12 Hours | 0.0 (12.68) | -3.3 (6.42) | -6.0 (13.06)
  Diastolic Blood Pressure- Change at 24 Hours | -0.5 (7.34) | -5.1 (5.56) | -11.4 (10.14)
  Diastolic Blood Pressure- Change at 8 Days | -3.0 (6.72) | -5.0 (9.55) | -7.6 (7.37)

5. Primary Outcome: Change From Baseline in Heart Rate at 0.5, 1, 1.5, 2.5, 3.5, 4.5, 5.5, 6.5, 9, 12, and 24 Hours, and Day 8 Post Dose
Description: as for outcome 1
Time Frame: Baseline and 0.5, 1, 1.5, 2.5, 3.5, 4.5, 5.5, 6.5, 9, 12, and 24 hours, and Day 8 post dose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Regimen 1 Conivaptan 12.5 mg | Regimen 2 Conivaptan 25 mg | Regimen 3 Placebo
Number analyzed (Participants) | 6 | 9 | 5
bpm
  Baseline | 69.0 (19.30) | 77.3 (22.86) | 72.0 (25.52)
  Change at 0.5 Hours | 0.7 (8.33) | -6.0 (11.88) | -2.0 (8.22)
  Change at 1 Hour | 3.0 (7.92) | -5.4 (9.25) | -2.4 (7.30)
  Change at 1.5 Hours | 2.3 (8.66) | -4.0 (9.73) | -3.2 (8.29)
  Change at 2.5 Hours | -0.3 (3.27) | -8.6 (11.17) | 0.4 (9.10)
  Change at 3.5 Hours | 1.3 (7.66) | -1.4 (14.34) | 2.8 (7.56)
  Change at 4.5 Hours | 3.3 (5.65) | -1.2 (15.81) | 4.0 (7.35)
  Change at 5.5 Hours | 4.3 (5.35) | -2.9 (14.14) | 3.6 (5.18)
  Change at 6.5 Hours | 8.0 (4.56) | -4.0 (13.08) | 3.4 (7.23)
  Change at 9 Hours | 4.8 (10.21) | -0.9 (12.32) | 1.8 (11.48)
  Change at 12 Hours | 1.8 (8.84) | 9.0 (21.46) | 3.8 (15.16)
  Change at 24 Hours | 1.2 (6.01) | 2.7 (17.00) | 3.6 (7.37)
  Change at 8 Days | 0.7 (10.31) | -7.1 (20.87) | -0.8 (9.18)

6. Secondary Outcome: Change From Baseline in Serum Sodium Levels at 0.5, 1, 2.5, 4, 6.5, 9, 12, and 24 Hours and on Day 8 Post Dose
Description: Baseline serum sodium value is the last measurement prior to dosing.
  Change from baseline is calculated as time point minus baseline.
Time Frame: Baseline and 0.5, 1, 2.5, 4, 6.5, 9, 12, and 24 hours and on Day 8 post dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | Regimen 1 Conivaptan 12.5 mg | Regimen 2 Conivaptan 25 mg | Regimen 3 Placebo
Number analyzed (Participants) | 6 | 9 | 5
mEq/L
  Baseline (N= 6; 9; 5) | 137.3 (3.08) | 137.1 (2.80) | 131.2 (6.30)
  Change at 0.5 Hours (N= 6; 9; 5) | -1.3 (3.01) | -1.1 (2.71) | -0.8 (1.64)
  Change at 1 Hour (N= 6; 9; 5) | -0.3 (3.72) | 0.9 (2.80) | -1.8 (1.30)
  Change at 2.5 Hours (N= 6; 9; 5) | 1.8 (2.56) | 0.2 (1.72) | 0.0 (3.61)
  Change at 4 Hours (N= 6; 9; 5) | -2.2 (5.19) | -1.0 (1.87) | -3.6 (1.67)
  Change at 6.5 Hours (N= 6; 9; 5) | -1.2 (2.32) | 1.3 (4.33) | -2.4 (2.07)
  Change at 9 Hours (N= 5; 9; 5) | -2.6 (3.05) | 0.8 (3.46) | -2.4 (2.97)
  Change at 12 Hours (N= 6; 9; 5) | -3.7 (2.66) | 0.1 (3.06) | -2.2 (2.28)
  Change at 24 Hours (N= 6; 9; 5) | -1.5 (2.88) | 0.1 (1.76) | -2.0 (3.16)
  Change at 8 Days (N= 6; 9; 5) | -2.3 (3.20) | 0.1 (3.59) | 2.0 (1.00)

ADVERSE EVENTS:
Description: Treatment-Emergent Adverse Event (TEAE) is an event that occurred after the first dose of study drug through 24 hours after the last dose of study drug.
Arm/Group | Regimen 1 Conivaptan 12.5 mg | Regimen 2 Conivaptan 25 mg | Regimen 3 Placebo
Serious Adverse Events (participants affected / at risk) | 0/6 | 2/9 | 0/5
Other Adverse Events (participants affected / at risk) | 1/6 | 6/9 | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Regimen 1 Conivaptan 12.5 mg (N=6) | Regimen 2 Conivaptan 25 mg (N=9) | Regimen 3 Placebo (N=5)
Atrial tachycardia (Cardiac disorders) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Regimen 1 Conivaptan 12.5 mg (N=6) | Regimen 2 Conivaptan 25 mg (N=9) | Regimen 3 Placebo (N=5)
Atrial flutter (Cardiac disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Polydipsia (Metabolism and nutrition disorders) | 0 | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Phlebitis (Vascular disorders) | 0 | 2 | 0

LIMITATIONS AND CAVEATS:
Company makes no warranties or representations of any kind as to the posting, expressed or implied, including warranties of merchantability and fitness for a particular purpose, and shall not be liable for any damages.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated from the Study. Sponsor must receive the manuscript 60 days prior to publication to ensure that no confidential information of Sponsor is included in the document. Sponsor may delay the publication for an additional 60 days to seek patent protection.